CLINICAL TRIAL: NCT02083640
Title: A Phase 1, Open-Label, 6 Sequence, 3 Period, Crossover Study Of Palbociclib (PD-0332991) In Healthy Volunteers To Estimate The Relative Bioavailability Of 3 Palbociclib Formulations
Brief Title: Relative Bioavailability For Palbociclib Formulations
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: A5481040
Record Dates: First submitted 2014-03-07; First posted 2014-03-11 (Estimated); Last update posted 2014-06-04 (Estimated); Status verified 2014-06

CONDITIONS: Healthy
Keywords: healthy volunteer; bioavailability; palbociclib; formulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Treatment A (Reference) (Other)
  Interventions: Drug: Palbociclib Formulation Reference
- Treatment B (Test) (Other)
  Interventions: Drug: Palbociclib Formulation Test
- Treatment C (Test) (Other)
  Interventions: Drug: Palbociclib Formulation Test

INTERVENTIONS:
Drug: Palbociclib Formulation Reference — 125 mg single dose of palbociclib formulation with 16 micrometer API particle size and dissolution level 1, which is representative of the intended commercial hard gelatin capsule.
  Arms: Treatment A (Reference)
Drug: Palbociclib Formulation Test — 125 mg single dose of palbociclib formulation with 41 micrometer API particle size and dissolution level 1
  Arms: Treatment B (Test)
Drug: Palbociclib Formulation Test — 125 mg single dose of palbociclib formulation with 16 micrometer API particle size and dissolution level 2
  Arms: Treatment C (Test)

SUMMARY:
This study is to assess the relative bioavailability of palbociclib hard gelatin capsule formulation (API 41 micrometer and dissolution Level 1) and palbociclib hard gelatin capsule formulation (API 16 micrometer and dissolution Level 2) compared to the palbociclib hard gelatin capsule formulation (API 16 micrometer and dissolution Level 1) after single 125 mg oral doses under fed conditions in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects and/or female subjects with no physical possibility of getting pregnant.
* Evidence of a personally signed and dated informed consent document indicating that the subject (or a legal representative) has been informed of all pertinent aspects of the study.
* Subjects who are willing and able to comply with all scheduled visits, treatment plan, laboratory tests, and other study procedures.

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease.
* Any condition possibly affecting drug absorption (eg, gastrectomy).
* A positive urine drug screen.
* History of regular alcohol consumption exceeding 7 drinks/week for females or 14 drinks/week for males (1 drink = 5 ounces (150 mL) of wine or 12 ounces (360 mL) of beer or 1.5 ounces (45 mL) of hard liquor) within 6 months of Screening.
* Treatment with an investigational drug within 30 days (or as determined by the local requirement, whichever is longer) preceding the first dose of study medication.
* Pregnant females; breastfeeding females; females with physical possibility of getting pregnant .

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2014-03; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Area Under the Curve From Time Zero to Extrapolated Infinite Time [AUC (0 - 8)] | 6 days
  AUC (0 - 8)= Area under the plasma concentration versus time curve (AUC) from time zero (pre-dose) to extrapolated infinite time (0 - 8). It is obtained from AUC (0 - t) plus AUC (t - 8).
Maximum Observed Plasma Concentration (Cmax) | 6 days

SECONDARY OUTCOMES:
Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClast) | 6 days
  Area under the plasma concentration time-curve from zero to the last measured concentration (AUClast)
Apparent Oral Clearance (CL/F) | 6 days
  Clearance of a drug is a measure of the rate at which a drug is metabolized or eliminated by normal biological processes. Clearance obtained after oral dose (apparent oral clearance) is influenced by the fraction of the dose absorbed. Clearance was estimated from population pharmacokinetic (PK) modeling. Drug clearance is a quantitative measure of the rate at which a drug substance is removed from the blood.
Time to Reach Maximum Observed Plasma Concentration (Tmax) | 2 Days
Apparent Volume of Distribution (Vz/F) | 6 days
  Volume of distribution is defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired plasma concentration of a drug. Apparent volume of distribution after oral dose (Vz/F) is influenced by the fraction absorbed.
Plasma Decay Half-Life (t1/2) | 6 days
  Plasma decay half-life is the time measured for the plasma concentration to decrease by one half.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, New Haven, Connecticut, United States

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A5481040&StudyName=Relative%20Bioavailability%20For%20Palbociclib%20Formulations